CLINICAL TRIAL: NCT01123161
Title: Phase 2/3 Study of Intravenous Thrombolysis and Hypothermia for Acute Treatment of Ischemic Stroke
Brief Title: The Intravascular Cooling in the Treatment of Stroke 2/3 Trial
Acronym: ICTuS2/3
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: The ICTuS 2 portion of the trial has been halted and data will be analyzed.
Sponsor: University of California, San Diego (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Patrick Lyden, Principal Investigator, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: ICTuS2/3; P50NS044148 (NIH); P50NS044227 (NIH)
Record Dates: First submitted 2010-04-27; First posted 2010-05-14 (Estimated); Results first posted 2017-04-05 (Actual); Last update posted 2017-04-05 (Actual); Status verified 2017-02

CONDITIONS: Stroke, Acute
Keywords: Hypothermia; Molecular Mechanisms of Pharmacological Action; Cerebral Infarction; Hematologic Agents; Stroke; Nervous System Diseases; Vascular Diseases; Tissue Plasminogen Activator; Central Nervous System Diseases; Fibrinolytic Agents; Cardiovascular Agents; Body Temperature Changes; Brain Diseases; Cerebrovascular Disorders; Pharmacologic Actions; Signs and Symptoms; Fibrin Modulating Agents; Therapeutic Uses; Brain Ischemia; Cardiovascular Diseases; Brain Infarction; Plasminogen; cooling; tPA; thrombolysis
MeSH Terms: conditions — Stroke; Hypothermia; Cerebral Infarction; Nervous System Diseases; Vascular Diseases; Central Nervous System Diseases; Body Temperature Changes; Brain Diseases; Cerebrovascular Disorders; Signs and Symptoms; Brain Ischemia; Cardiovascular Diseases; Brain Infarction | interventions — Cool-Down Exercise

STUDY DESIGN:
Intervention Model Description: Randomized to normothermia or hypothermia
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group1: IV t-PA and normothermia (Active Comparator): IV tpa and normothermia
  Interventions: Drug: Group1: IV t-PA and normothermia
- Group 2 : IV t-PA and hypothermia and anti-shivering treatment (Active Comparator): IV tpa and hypothermia and anti-shivering treatment
  Interventions: Device: hypothermia and anti-shivering treatment

INTERVENTIONS:
Device: hypothermia and anti-shivering treatment — Hypothermia is induced using the Celsius Control™ System. Shivering is treated with buspirone, meperidine and surface warming
  Other Names: cooling
  Arms: Group 2 : IV t-PA and hypothermia and anti-shivering treatment
Drug: Group1: IV t-PA and normothermia — Group 1 will t-PA as standard of care and normothermia
  Arms: Group1: IV t-PA and normothermia

SUMMARY:
The purpose of this trial is to determine whether the combination of thrombolysis and hypothermia is superior to thrombolysis alone for the treatment of acute ischemic stroke.

DETAILED DESCRIPTION:
A stroke is usually caused by a blockage in one of the arteries that carries blood to the brain. Research has shown that tissue plasminogen activator (tPA)-a naturally occurring protein that opens blocked arteries by dissolving blood clots - activates the body's ability to dissolve recently formed blood clots and reduces or prevents the brain damage caused by a stroke.

The Food and Drug Administration (FDA) has approved the use of tPA for people having a stroke when taken within 3 hours of stroke onset.

Researchers believe that a lower body temperature (hypothermia) may be beneficial while a stroke is happening because hypothermia may prevent further brain injury, or may make the stroke less damaging.

Patients will receive a standard stroke evaluation, which includes blood tests, a computed tomography (CT) scan, complete physical and neurological examinations, and an electrocardiogram (EKG) to determine eligibility for the study.

There are two study groups - tPA alone or tPA with cooling (hypothermia). Participants will be randomly assigned to one of the two study groups. Length of participation (including observation after the patient leaves the hospital) is 90 days.

This study is part of the Specialized Program of Translational Research in Acute Stroke (SPOTRIAS), which allows researchers to enhance and initiate translational research that ultimately will benefit stroke patients by treating more patients in less than 2 hours, and finding ways to treat additional patients later.

ELIGIBILITY:
Inclusion Criteria:

1. Age 22 to 82 years old inclusive
2. Patient receiving IV rt-PA using standard guidelines
3. NIHSS score ≥ 7 and ≤ 20 (right hemisphere) or ≥ 7 and ≤ 24 (left hemisphere) at the time of randomization
4. Pre-stroke mRS 0-1
5. Able to begin endovascular phase of hypothermia within 2 hours of tPA completion
6. Written Informed Consent, signed and dated by the patient (or patient's authorized representative)

Exclusion Criteria:

1. Etiology other than ischemic stroke
2. Item 1a on NIHSS > 1 at the time of randomization
3. Clinical symptoms consistent with brainstem or cerebellar stroke
4. Classic lacunar syndrome with imaging confirmation of small deep ischemia, but randomization will not be delayed for neuroimaging other than initial scan to exclude hemorrhage
5. Known contraindications to hypothermia, such as known hematologic dyscrasias that affect thrombosis (cryoglobulinemia, Sickle cell disease, serum cold agglutinins), or vasospastic disorders such as Raynaud's or thromboangiitis obliterans
6. Known co-morbid conditions that are likely to complicate therapy in the opinion of the investigator, e.g., i. Heart failure (NYHA class III and IV)* ii. Uncompensated arrhythmia iii. Severe Liver disease iv. History of pelvic or abdominal mass likely to compress inferior vena cava v. IVC filters vi. HIV positive vii. Clinically active hypo or hyperthyroidism viii. Renal insufficiency likely to impair meperidine clearance ix. Chronic ethanol abuse x. History of HIT (heparin induced thrombocytopenia)
7. Pregnancy (All women of child-bearing potential must have a negative pregnancy test, urine or blood, prior to therapy.)
8. Medical conditions likely to interfere with patient assessment.
9. Known allergy to meperidine or buspirone
10. Currently taking or used within previous 14 days MAO-I class of medication.
11. Life expectancy < 6 months
12. Not likely to be available for long-term follow-up
13. Use, or planned use, of intra-arterial thrombolysis, mechanical clot removal, or other experimental or approved acute therapy for this stroke event
14. Chest radiograph or clinical presentation suggestive of pneumonia or clinically significant pulmonary edema at baseline.
15. Temperature upon admission greater than or equal to 38°C

Ages: 22 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2010-06; Primary Completion 2015-01 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick D. Lyden, MD, Principal Investigator — Cedars-Sinai Medical Center; Thomas M. Hemmen, MD, PhD, Study Director — University of California, San Diego; James C. Grotta, MD, Study Director — The University of Texas Health Science Center, Houston
Locations (31):
- United States (29):
  - University of Alabama Hospital, Birmingham, Alabama
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - University of California San Diego Health System, San Diego, California
  - Scripps Mercy Medical Center, San Diego, California
  - University of Colorado Hospital, Aurora, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Gulf Coast Medical Center, Fort Myers, Florida
  - University of Florida, Gainesville, Florida
  - University of Miami, Jackson Memorial Hospital, Miami, Florida
  - Intercoastal Medical Group, Sarasota, Florida
  - St. Joseph's Hospital, Tampa, Florida
  - Alexian Brothers Medical Center, Elk Grove Village, Illinois
  - Parkview Hospital, Fort Wayne, Indiana
  - Ruan Neurology Clinic and Research Center, Des Moines, Iowa
  - University of Louisville, Louisville, Kentucky
  - Henry Ford Health System, Detroit, Michigan
  - Michigan State University, East Lansing, Michigan
  - North Memorial Medical Center, Robbinsdale, Minnesota
  - Saint Louis University Medical Center, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - University of Toledo Medical Center, Toledo, Ohio
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Lehigh Valley Health Network, Allentown, Pennsylvania
  - Seton Medical Center Austin, Austin, Texas
  - UT Southwestern, Dallas, Texas
  - University of Texas Health Science Center, Houston, Texas
- Medical University Innsbruck, Innsbruck, Austria
- CHUV, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lyden PD, Allgren RL, Ng K, Akins P, Meyer B, Al-Sanani F, Lutsep H, Dobak J, Matsubara BS, Zivin J. Intravascular Cooling in the Treatment of Stroke (ICTuS): early clinical experience. J Stroke Cerebrovasc Dis. 2005 May-Jun;14(3):107-14. doi: 10.1016/j.jstrokecerebrovasdis.2005.01.001. PMID 17904009
- [Background] Hemmen TM, Raman R, Guluma KZ, Meyer BC, Gomes JA, Cruz-Flores S, Wijman CA, Rapp KS, Grotta JC, Lyden PD; ICTuS-L Investigators. Intravenous thrombolysis plus hypothermia for acute treatment of ischemic stroke (ICTuS-L): final results. Stroke. 2010 Oct;41(10):2265-70. doi: 10.1161/STROKEAHA.110.592295. Epub 2010 Aug 19. PMID 20724711
- [Background] Lyden P, Ernstrom K, Raman R. Determinants of Pneumonia Risk During Endovascular Hypothermia. Ther Hypothermia Temp Manag. 2013 Mar;3(1):24-27. doi: 10.1089/ther.2012.0021. PMID 23667781
- [Background] Lyden P, Ernstrom K, Cruz-Flores S, Gomes J, Grotta J, Mullin A, Rapp K, Raman R, Wijman C, Hemmen T. Determinants of effective cooling during endovascular hypothermia. Neurocrit Care. 2012 Jun;16(3):413-20. doi: 10.1007/s12028-012-9688-y. PMID 22466971
- [Background] Guluma KZ, Liu L, Hemmen TM, Acharya AB, Rapp KS, Raman R, Lyden PD. Therapeutic hypothermia is associated with a decrease in urine output in acute stroke patients. Resuscitation. 2010 Dec;81(12):1642-7. doi: 10.1016/j.resuscitation.2010.08.003. PMID 20817376
- [Background] Guluma KZ, Hemmen TM, Olsen SE, Rapp KS, Lyden PD. A trial of therapeutic hypothermia via endovascular approach in awake patients with acute ischemic stroke: methodology. Acad Emerg Med. 2006 Aug;13(8):820-7. doi: 10.1197/j.aem.2006.03.559. Epub 2006 Jun 9. PMID 16766740
- [Derived] Lyden P, Hemmen T, Grotta J, Rapp K, Ernstrom K, Rzesiewicz T, Parker S, Concha M, Hussain S, Agarwal S, Meyer B, Jurf J, Altafullah I, Raman R; Collaborators. Results of the ICTuS 2 Trial (Intravascular Cooling in the Treatment of Stroke 2). Stroke. 2016 Dec;47(12):2888-2895. doi: 10.1161/STROKEAHA.116.014200. Epub 2016 Nov 10. PMID 27834742

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 2 : IV t-PA and Hypothermia and Anti-shivering Treatment: IV tpa and hypothermia and anti-shivering treatment
  hypothermia: Hypothermia is induced using the Celsius Control™ System. Shivering is treated with buspirone, meperidine, and surface warming.
Period: Overall Study
Arm/Group | Group1: IV t-PA and Normothermia | Group 2 : IV t-PA and Hypothermia and Anti-shivering Treatment
Started | 57 | 63
Completed | 55 | 63
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Patients enrolled and randomized
Groups:
- Total: Total of all reporting groups
Arm/Group | Group1: IV t-PA and Normothermia | Group 2 : IV t-PA and Hypothermia and Anti-shivering Treatment | Total
Number analyzed (Participants) | 57 | 63 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.5 (11.1) | 65.5 (10.3) | 66.4 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 29 | 51
  Male | 35 | 34 | 69
Baseline NIHSS [Mean (Standard Deviation); unit: points] — The NIHSS measures neurological deficit. Scores range from 0 (best) to 42 (worst). Between 0 and 42 higher scores reflect progressively worse neurological deficit.
  points | 14.5 (4.9) | 14.1 (4.8) | 14.3 (4.8)
Baseline temperature [Mean (Standard Deviation); unit: degrees (C)] | 36.4 (0.50) | 36.6 (0.46) | 36.5 (0.48)

OUTCOME MEASURES:

1. Primary Outcome: The Primary Outcome is the Proportion of Patients Achieving a Favorable Outcome Defined as Modified Rankin Scale Score of 0 or 1, Assessed 90 Days After Treatment.
Description: Modified Rankin describes disability: 0 is free of any disability or symptoms, 6 is death, and higher grades between 0 and 6 reflect progressively greater disability
Time Frame: 90 days
Population: Intention to Treat Population
Measure: Number; unit: participants
Groups:
- Group 2 : IV t-PA and Hypothermia: IV tpa and hypothermia
  hypothermia: Hypothermia is induced using the Celsius Control™ System
Arm/Group | Group1: IV t-PA and Normothermia | Group 2 : IV t-PA and Hypothermia
Number analyzed (Participants) | 55 | 63
participants | 21 | 21

2. Primary Outcome: Incidence of Any Intracranial Hemorrhage (ICH) Within 48 Hours of Stroke Onset
Description: Incidence (number) of any intracranial hemorrhage (ICH) (whether or not symptomatic) within 48 hours of stroke onset will be presented by treatment group and overall.
Time Frame: 48 hours
Population: Intention to treat patients with imaging obtained 36 to 48 hours after treatment
Measure: Number; unit: participants
Arm/Group | Group1: IV t-PA and Normothermia | Group 2 : IV t-PA and Hypothermia and Anti-shivering Treatment
Number analyzed (Participants) | 57 | 63
participants | 13 | 9

3. Primary Outcome: Incidence of Any Symptomatic Intracranial Hemorrhage (sICH) Within 48 Hours of Stroke Onset
Description: Incidence (number) of Symptomatic ICH (sICH) within 48 hours of stroke onset will be presented by treatment group and overall. Patients with neuroworsening (4 or more point increase in NIHSS , or a decline in the NIHSS consciousness item 1A score of more than 1 point, or a motor deterioration lasting more than 8 hours, all not due to iatrogenic cause) and hemorrhage seen on brain images in whom the investigator attributes the clinical change to the hemorrhage.
Time Frame: 48 hours
Population: ITT patients in whom a brain image was obtained 36 yo 48 hours after treatment
Measure: Number; unit: participants
Arm/Group | Group1: IV t-PA and Normothermia | Group 2 : IV t-PA and Hypothermia and Anti-shivering Treatment
Number analyzed (Participants) | 57 | 63
participants | 2 | 1

4. Primary Outcome: Incidence of Pneumonia
Description: Number subjects diagnosed with pneumonia according to CDC criteria will be presented by treatment group and overall, regardless of seriousness
Time Frame: 7 days or discharge whichever comes first
Population: ITT population
Measure: Number; unit: participants
Arm/Group | Group1: IV t-PA and Normothermia | Group 2 : IV t-PA and Hypothermia and Anti-shivering Treatment
Number analyzed (Participants) | 57 | 63
participants | 6 | 12

5. Primary Outcome: 90 Day Mortality
Description: Mortality prior to the 90-day evaluation.
Time Frame: 90 days
Population: ITT population
Measure: Number; unit: participants
Arm/Group | Group1: IV t-PA and Normothermia | Group 2 : IV t-PA and Hypothermia and Anti-shivering Treatment
Number analyzed (Participants) | 57 | 63
participants | 5 | 10

6. Secondary Outcome: The Barthel Index Measure of Activities of Daily Living;
Description: The Barthel index measures independence in activities of daily living from 0 (worst) to 100 (best) in 5 point increments. Higher scores between 0 and 100 reflect progressively greater levels of independence. Scores were dichotomized at 90 so that a score of 95 or 100 was considered a successful treatment.
Time Frame: 90 days
Population: The intention to treat population with a 90-day Barthel index available was used, therefore the numbers are fewer than in the total population.
Measure: Number; unit: participants
Groups:
- Group 2 : IV t-PA and Hypothermia and Anti-shivering Treatment: IV tpa and hypothermia
  hypothermia: Hypothermia is induced using the Celsius Control™ System. Shivering treatment includes buspirone, meperidine, and surface warming.
Arm/Group | Group1: IV t-PA and Normothermia | Group 2 : IV t-PA and Hypothermia and Anti-shivering Treatment
Number analyzed (Participants) | 46 | 49
participants | 25 | 24

7. Secondary Outcome: NIHSS Scores at 90 Days
Description: The National Institutes of Health Stroke Scale (NIHSS) is used to quantify neurological deficit. The scale ranges from 0 (best) to 42 points (worst). Between scores of 0 to 42, higher values reflect progressively greater deficit.
Time Frame: 90 days
Population: Intention to treat patients with an available 90-day NIHSS values therefore the total numbers available are fewer than the total ITT population.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group1: IV t-PA and Normothermia | Group 2 : IV t-PA and Hypothermia and Anti-shivering Treatment
Number analyzed (Participants) | 44 | 43
units on a scale | 6.1 (6.6) | 4.8 (5.4)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for 7 days or discharge whichever came first. Serious adverse events were collected for 90 days.
Description: Adverse events and Other (not including serious) events are summarized by system organ class, rather than Adverse Event Terms, due to the small number of subjects and infrequency of adverse events.
Groups:
- Group 2 : IV t-PA and Hypothermia and Anti-shivering Treatment: IV tpa and hypothermia and anti-shivering treatment
  hypothermia: Hypothermia is induced using the Celsius Control™ System. Shivering is treated with buspirone, meperidine and surface warming.
Arm/Group | Group1: IV t-PA and Normothermia | Group 2 : IV t-PA and Hypothermia and Anti-shivering Treatment
Serious Adverse Events (participants affected / at risk) | 20/57 | 26/63
Other Adverse Events (participants affected / at risk) | 53/57 | 63/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group1: IV t-PA and Normothermia (N=57) | Group 2 : IV t-PA and Hypothermia and Anti-shivering Treatment (N=63)
Cardiac Disorders (Cardiac disorders) | 3 (3) | 2 (2) — arrest, CHF, CAD, cardiomyopathy
Infections (Infections and infestations) | 0 (0) | 4 (4) — bacteremia, sepsis, shock
injury (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) — contusion, muscle injury, pelvic fracture
Metabolism (Metabolism and nutrition disorders) | 0 (0) | 2 (2) — dehydration, metabolic acidosis
muskuloskeletal (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — ankle fracture
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) — metastases to meninges
Nervous System Disorders (Nervous system disorders) | 13 (17) | 13 (13) — agitation, herniation, oedema, carotid artery stenosis, cerebral hemorrhage, confusional state, ICH, sedation, stroke in evolution
psychiatric disorders (Psychiatric disorders) | 0 (0) | 1 (1) — delerium
renal (Renal and urinary disorders) | 0 (0) | 1 (1) — renal failure
Respiratory (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 9 (10) — ARDs, respiratory failure, pneumonia, PE, resp distress, resp depression, resp failure
vascular (Vascular disorders) | 3 (4) | 1 (1) — Arterial rupture, deep vein thrombosis, Hemorrhage, or hypotension
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group1: IV t-PA and Normothermia (N=57) | Group 2 : IV t-PA and Hypothermia and Anti-shivering Treatment (N=63)
Blood and lymphatic (Blood and lymphatic system disorders) | 7 (7) | 4 (4) — Total AEs
Cardiac (Cardiac disorders) | 15 (16) | 19 (33)
Endocrine (Endocrine disorders) | 0 (0) | 6 (6)
Eye (Eye disorders) | 2 (2) | 2 (2)
GI (Gastrointestinal disorders) | 23 (30) | 36 (50)
General (General disorders) | 17 (21) | 34 (38)
immune (Immune system disorders) | 1 (1) | 2 (2)
Infection (Infections and infestations) | 10 (11) | 14 (14)
injury (Injury, poisoning and procedural complications) | 6 (6) | 7 (7)
investigations (Investigations) | 34 (83) | 52 (139)
Metabolism (Metabolism and nutrition disorders) | 6 (6) | 11 (11)
Muskuloskeletal (Musculoskeletal and connective tissue disorders) | 7 (8) | 11 (12)
Neoplasms (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Nervous Systen (Nervous system disorders) | 33 (54) | 37 (46)
Psychiatric (Psychiatric disorders) | 8 (8) | 8 (8)
Renal (Renal and urinary disorders) | 6 (6) | 5 (6)
Reproductive (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Respiratory (Respiratory, thoracic and mediastinal disorders) | 15 (21) | 31 (44)
Skin (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Vascular (Vascular disorders) | 19 (23) | 28 (33)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No